CLINICAL TRIAL: NCT03662919
Title: PERFUSE - One-year Persistence to Treatment of Patients Receiving Flixabi or Imraldi: a French Cohort Study
Brief Title: One-year Persistence to Treatment of Participants Receiving Flixabi or Imraldi: a French Cohort Study
Acronym: PERFUSE
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: FRA-FLX-17-11226; 2017-A03220-53 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Crohn's Disease; Colitis, Ulcerative
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Crohn Disease; Colitis, Ulcerative | interventions — Infliximab; Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Flixabi: Infliximab naive participants or participants who were previously treated with other infliximab biologics will receive Flixabi (infliximab) as prescribed by physician according to the local prescribing procedures.
  Interventions: Drug: Infliximab
- Imraldi: Adalimumab naive participants or participants who were previously treated with other adalimumab biosimilars will receive Imraldi (adalimumab) as prescribed by physician according to the local prescribing procedures.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Infliximab — Administered as specified in the treatment arm.
  Other Names: Flixabi
  Groups: Flixabi
Drug: Adalimumab — Administered as specified in the treatment arm.
  Other Names: Imraldi
  Groups: Imraldi

SUMMARY:
A study to describe the one-year persistence in participants treated by Flixabi (infliximab) or Imraldi (Adalimumab) as prescribed by the physician for each of the 5 following indications: Rheumatoid Arthritis (RA), Ankylosing Spondylitis (AS), Psoriatic Arthritis (PsA), Crohn's Disease (CD) [adults and children] and Ulcerative Colitis (UC) [adults for both treatments and children only for Flixabi].

ELIGIBILITY:
Inclusion/ Exclusion Criteria

Key Inclusion Criteria:

* Adult participant (18 years and over)

  * treated for one of the following conditions: RA, AS, PsA, CD, UC.
  * either active substance naïve or treated with the originator or another biosimilar at baseline.
  * for whom the treating physician has decided to treat by (naïve) or switch from originator or another biosimilar to Flixabi or Imraldi.
  * participants who had initiated Flixabi or Imraldi at most 12 months before the baseline will also be included in the cohort.
* Paediatric participants (6-17 years):

  * treated for one of the following conditions: CD, UC.
  * either active substance naïve or treated with another biosimilar at baseline.
  * for whom the treating physician has decided to treat by (naïve) or switch to Flixabi (for both indications) or Imraldi (only for Crohn's disease).
  * participants who had initiated Flixabi or Imraldi at most 12 months before the baseline will also be included in the cohort.

Key Exclusion Criteria:

* Participant treated for psoriasis.
* Participant who are not to be followed up in the same investigator site for 2 years after baseline.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants either infliximab naïve or switched from Remicade or CT-P13 to Flixabi who are treated with Flixabi, and either adalimumab naïve or switched from Humira or other adalimumab biosimilars to Imraldi who are treated with Imraldi, for RA, AS, PsA, CD, and UC as prescribed by the physician in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 2274 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who are Still Treated with Either Flixabi or Imraldi at 12 Months | Up to 12 months
  Percentage of participants, either infliximab naïve or switched from Remicade or CT-P13 to Flixabi, who are still treated with Flixabi, and either adalimumab naïve or switched from Humira or other adalimumab biosimilars to Imraldi, who are still treated with Imraldi, at 12 months for RA, AS, PsA, CD (adults and children), and UC (adults for both treatments and children only for Flixabi) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (60):
- France (60):
  - Research Site, Caluire-et-Cuire, Auvergne-Rhône-Alpes
  - Research Site 1, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Research Site, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Research Site, Lyon, Auvergne-Rhône-Alpes
  - Research Site 1, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Research Site, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Research Site, Saint-Etienne, Auvergne-Rhône-Alpes
  - Research Site, Dijon, Bourgogne-Franche-Comté
  - Research Site 1, Brest, Brittany Region
  - Research Site, Brest, Brittany Region
  - Research Site, Rennes, Brittany Region
  - Research Site, Chambray-lès-Tours, Centre-Val de Loire
  - Research Site, Orléans, Centre-Val de Loire
  - Research Site, Reims, Grand Est
  - Research Site, Strasbourg, Grand Est
  - Research Site 1, Vandœuvre-lès-Nancy, Grand Est
  - Research Site, Vandœuvre-lès-Nancy, Grand Est
  - Research Site, Amiens, Hauts-de-France
  - Research Site 1, Lille, Hauts-de-France
  - Research Site, Lille, Hauts-de-France
  - Research Site, Caen, Normandy
  - Research Site, Rouen, Normandy
  - Research Site, Bayonne, Nouvelle-Aquitaine
  - Research Site, Bordeaux, Nouvelle-Aquitaine
  - Research Site 1, La Rochelle, Nouvelle-Aquitaine
  - Research Site 2, La Rochelle, Nouvelle-Aquitaine
  - Research Site, La Rochelle, Nouvelle-Aquitaine
  - Research Site, Limoges, Nouvelle-Aquitaine
  - Research Site 1, Montpellier, Occitanie
  - Research Site, Montpellier, Occitanie
  - Research Site 1, Nîmes, Occitanie
  - Research Site, Nîmes, Occitanie
  - Research Site 1, Toulouse, Occitanie
  - Research Site, Toulouse, Occitanie
  - Research Site, Angers, Pays de la Loire Region
  - Research Site 1, Nantes, Pays de la Loire Region
  - Research Site, Nantes, Pays de la Loire Region
  - Research Site, Cannes, Provence-Alpes-Côte d'Azur Region
  - Research Site, La Crau, Provence-Alpes-Côte d'Azur Region
  - Research Site 1, Marseille, Provence-Alpes-Côte d'Azur Region
  - Research Site, Marseille, Provence-Alpes-Côte d'Azur Region
  - Research Site, Nice, Provence-Alpes-Côte d'Azur Region
  - Research Site, Toulon, Provence-Alpes-Côte d'Azur Region
  - Research Site 1, Bobigny, Île-de-France Region
  - Research Site, Bobigny, Île-de-France Region
  - Research Site, Clichy, Île-de-France Region
  - Research Site, Colombes, Île-de-France Region
  - Research Site, Créteil, Île-de-France Region
  - Research Site, Le Kremlin-Bicêtre, Île-de-France Region
  - Research Site 10, Paris, Île-de-France Region
  - Research Site 1, Paris, Île-de-France Region
  - Research Site 2, Paris, Île-de-France Region
  - Research Site 3, Paris, Île-de-France Region
  - Research Site 4, Paris, Île-de-France Region
  - Research Site 5, Paris, Île-de-France Region
  - Research Site 6, Paris, Île-de-France Region
  - Research Site 7, Paris, Île-de-France Region
  - Research Site 8, Paris, Île-de-France Region
  - Research Site 9, Paris, Île-de-France Region
  - Research Site, Paris, Île-de-France Region

REFERENCES:
- [Derived] Fautrel B, Bouhnik Y, Salliot C, Carbonnel F, Fumery M, Bernardeau C, Maugars Y, Flamant M, Coury F, Braithwaite B, Hateb S, Addison J; PERFUSE investigators. Real-World Evidence of Clinical Outcomes of the Use of the Adalimumab Biosimilar SB5 in Rheumatic and Gastrointestinal Immune-Mediated Inflammatory Diseases: 12-Month Data from the PERFUSE Study. Drugs Real World Outcomes. 2024 Dec;11(4):573-591. doi: 10.1007/s40801-024-00459-6. Epub 2024 Oct 10. PMID 39384685
- [Derived] Fautrel B, Bouhnik Y, Dieude P, Richette P, Dougados M, Freudensprung U, Brigui A, Addison J. Real-world evidence of the use of the infliximab biosimilar SB2: data from the PERFUSE study. Rheumatol Adv Pract. 2023 Apr 17;7(2):rkad031. doi: 10.1093/rap/rkad031. eCollection 2023. PMID 37122809
- [Derived] Martinez-Vinson C, Lemoine A, Bouhnik Y, Braithwaite B, Fohlen-Weill A, Addison J. PERFUSE: Non-Interventional Cohort Study of Patients Receiving Infliximab Biosimilar SB2: Results in Pediatric Patients. J Pediatr Gastroenterol Nutr. 2023 Apr 1;76(4):451-459. doi: 10.1097/MPG.0000000000003683. Epub 2022 Dec 16. PMID 36729422